CLINICAL TRIAL: NCT03066388
Title: Accuracy of Pulse Pressure Variations Measured by a Non Invasive Digital Device to Predict Fluid Responsiveness in Patients With Systemic Inflammatory Response Syndrome
Brief Title: Accuracy of Pulse Pressure Variations Measured by a Non Invasive Digital Device to Predict Fluid Responsiveness
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: insufficient inclusion rate
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2011_47; 2011-A01599-32 (Other: ID-RCB number)
Record Dates: First submitted 2016-11-09; First posted 2017-02-28 (Actual); Last update posted 2017-02-28 (Actual); Status verified 2017-02

CONDITIONS: Systemic Inflammatory Response Syndrome; Circulatory Failure; Mechanical Ventilation
Keywords: fluid; fluid responsiveness; pulse pressure; noninvasive monitoring; pulse pressure variations; volume expansion; SIRS; systemic inflammatory response syndrome
MeSH Terms: conditions — Systemic Inflammatory Response Syndrome; Shock

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pulse pressure variations (Experimental): Pulse pressure variations, stroke volume, systemic arterial pressure, heart rate, and respiratory rate are recorded immediately before and after volume expansion (VE), performed as a 30-minute infusion of 500 mL of 4% gelatin. Pulse pressure variations are obtained by noninvasive (ΔPPCNAP) and invasive (ΔPPART) devices.
  Interventions: Other: Pulse pressure variations

INTERVENTIONS:
Other: Pulse pressure variations — Stroke volume and, pulse pressure variations obtained by noninvasive (ΔPPCNAP) and invasive (ΔPPART) devices are recorded immediately before and after volume expansion (VE), performed as a 30-minute infusion of 500 mL of 4% gelatin.

SUMMARY:
It has been well established that only 40 to 60% of the patients hospitalized for inflammatory response syndrome (SIRS) positively respond to volume expansion (VE). The fluid responsiveness is usually estimated by assessing VE-induced change in stroke volume (SV). To guide prescriptions and possibly avoid deleterious effects of inappropriate VE, several clinical studies demonstrated that invasive dynamic indices based on heart-lung interactions permit an accurate prediction of the hemodynamic effects induced by VE.

Mechanical ventilation induces cyclic changes in intrathoracic and transpulmonary pressures that transiently affect venous return, right and left ventricular preload, resulting in pronounced cyclic changes in SV in preload-dependent, but not in preload-independent patients. These cyclic changes in SV can be evaluated by the cyclic changes in arterial pulse pressure. Several studies have shown that pulse pressure variation is able to predict fluid responsiveness in patients in the operating room and intensive care unit (ICU).

However, this technique requires percutaneous arterial catheterization, which is associated with several rare but serious complications (thrombosis, infections, pseudoaneurysm,hematoma, and bleeding).

A method for assessing noninvasive arterial blood pressure using an electropneumatic control loop was introduced by Penaz in 1973. Briefly, the blood volume in a finger is measured and kept constant by applying corresponding external pressure. The continuously changing external pressure needed to keep the volume constant directly corresponds to the arterial pressure and, therefore can be used as continuous measurement of arterial blood pressure. Numerous studies evaluating the accuracy of this technology, e.g., Finapres™ (Ohmeda Monitoring Systems, Englewood, CO), and more recently of the Infinity CNAP™ SmartPod (Dräger Medical AG & Co.KG, Lübeck, Germany).

The basic operating principle of the CNAP™ is similar to the Finapres™, but CNAP™ uses multiple control loops. It has recently been shown that CNAP provides real-time estimates of mean arterial blood pressure (MAP) comparable with those measured by an invasive intraarterial catheter system during general anaesthesia.

The accuracy of the measures and the respiratory variations in pulse pressure obtained with the CNAP system have not yet been studied in ICU.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients of the intensive care units of the Lille university-hospital.
* Age greater than or equal to 18.
* Patient insured
* Mechanical ventilation without spontaneous respiratory cycles
* Regular cardiac rhythm
* Prescription by the physician in charge of the patients of a 500 mL volume expansion in less than 30 minutes.
* Patients with sepsis with at least one sign of acute circulatory failure:

  * Tachycardia with heart rate> 100/min
  * systolic blood pressure <90mmHg or a decrease >40mmHg in previously hypertense patient
  * Oliguria <0.5ml/kg/hour for at least one hour
  * skin mottling

Exclusion Criteria:

* high-grade aortic insufficiency
* transthoracic echogenicity unsuitable for measuring the stroke volume by echo-Doppler
* Spontaneous breathing
* clinical or ultrasonographic evidence of pulmonary edema due to heart failure
* pregnancy
* abdominal compartment syndrome
* Irregular cardiac rhythm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2012-04; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
respiratory variations in noninvasive pulse pressure with respect to the response to fluid | during 30 minutes of the volume expansion

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien Preau, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Intensive Care Department, Salengro Hospital,CHRU, Lille, France

IPD SHARING:
Plan to Share IPD: No